CLINICAL TRIAL: NCT00354341
Title: An Open, Randomized, Multi-centre Trial to Investigate the Effect of Anemia Correction on Cardiac Structure and Function in Patients With Early Diabetic Nephropathy
Brief Title: (ACORD Study) - A Study of NeoRecormon (Epoetin Beta) in Patients With Early Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA16620
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (2):
- Group 1 (Early Epoetin Beta) (Experimental): Along with their standard treatment participants will receive epoetin beta at a starting dose of 2000 International Units (IU) subcutaneously (SC) once weekly to reach and maintain target hemoglobin (Hb) between 13 and 15 grams per deciliter (g/dL), for 15 months. Epoetin beta doses will be adjusted according to individual participant's Hb level. Standard treatment will be as per investigator discretion.
  Interventions: Drug: Epoetin beta
- Group 2 (No/Late Epoetin Beta) (Active Comparator): Participants will receive their standard treatment for 15 months but no treatment for anemia correction unless Hb level will be less than (<) 10.5 g/dL on 2 consecutive visits of 2 weeks interval or the Hb level will be <10 g/dL on a single determination. In such cases participants could receive epoetin beta at a starting dose of 2000 IU SC once weekly to reach and maintain a target Hb level of 10.5 to 11.5 g/dL. Standard treatment will be as per investigator discretion.
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta
  Other Names: NeoRecormon

SUMMARY:
This study will assess the effect of anemia correction with NeoRecormon on cardiac structure and function in patients with early diabetic nephropathy. The anticipated time on study treatment is 1-2 years and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* type 1 or type 2 diabetes;
* stable glycemic control for >=3 months;
* diabetic nephropathy.

Exclusion Criteria:

* women who are pregnant, breastfeeding, or unwilling to use a reliable contraceptive method;
* previous treatment with erythropoietin or other erythropoietic substance;
* nondiabetic renal disease, nephrotic syndrome;
* blood transfusion within the 3 months prior to enrollment;
* administration of any investigational drug within 30 days preceding the study start, and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2002-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebenhard Ritz, Prof. Dr., Principal Investigator — unaffliated
Locations (52):
- Linz, Austria
- São Paulo, Brazil
- Czechia (2):
  - Jihlava
  - Liberec
- Denmark (2):
  - Copenhagen
  - Roskilde
- Jyväskylä, Finland
- Germany (2):
  - Heidelberg
  - München
- Greece (6):
  - Alexandroupoli
  - Athens
  - Ioannina
  - Nikaia
  - Thessaloniki
  - Véria
- Hungary (4):
  - Budapest
  - Miskolc
  - Pécs
  - Szombathely
- Italy (8):
  - Ancona
  - Cagliari
  - Caserta
  - Cinisello Balsamo
  - Desio
  - Lecco
  - Messina
  - Milan
- Mexico (3):
  - Chihuahua City
  - Mexico City
  - Monterrey
- Poland (3):
  - Bialystok
  - Katowice
  - Radom
- Moscow, Russia
- Singapore, Singapore
- Spain (6):
  - A Coruña
  - Barakaldo
  - Barcelona
  - Galdakao
  - Madrid
  - Valencia
- Stockholm, Sweden
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Chon Buri
- United Kingdom (7):
  - Belfast
  - Cambridge
  - London
  - Middlesbrough
  - Salford
  - Sheffield
  - Wrexham

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Ritz E, Laville M, Bilous RW, O'Donoghue D, Scherhag A, Burger U, de Alvaro F; Anemia Correction in Diabetes Study Investigators. Target level for hemoglobin correction in patients with diabetes and CKD: primary results of the Anemia Correction in Diabetes (ACORD) Study. Am J Kidney Dis. 2007 Feb;49(2):194-207. doi: 10.1053/j.ajkd.2006.11.032. PMID 17261422

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Early Epoetin Beta): Along with their standard treatment participants received epoetin beta at a starting dose of 2000 International Units (IU) subcutaneously (SC) once weekly to reach and maintain target hemoglobin (Hb) between 13 and 15 grams per deciliter (g/dL), for 15 months. Epoetin beta doses were adjusted according to individual participant's Hb level. Standard treatment was as per investigator discretion.
- Group 2 (No/Late Epoetin Beta): Participants received their standard treatment for 15 months but no treatment for anemia correction unless Hb level was less than (<) 10.5 g/dL on 2 consecutive visits of 2 weeks interval or the Hb level was <10 g/dL on a single determination. In such cases participants could receive epoetin beta at a starting dose of 2000 IU SC once weekly to reach and maintain a target Hb level of 10.5 to 11.5 g/dL. Standard treatment was as per investigator discretion.
Period: Overall Study
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Started | 88 | 82
Completed | 85 | 75
Not Completed | 3 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 2
Not completed — Refused treatment | 1 | 2
Not completed — Failure to return | 0 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least one dose of study medication.
Groups:
- Group 1 (Early Epoetin Beta): Along with their standard treatment participants received epoetin beta at a starting dose of 2000 IU SC once weekly to reach and maintain target Hb between 13 and 15 g/dL, for 15 months. Epoetin beta doses were adjusted according to individual participant's Hb level. Standard treatment was as per investigator discretion.
- Group 2 (No/Late Epoetin Beta): Participants received their standard treatment for 15 months but no treatment for anemia correction unless Hb level was <10.5 g/dL on 2 consecutive visits of 2 weeks interval or the Hb level was <10 g/dL on a single determination. In such cases participants could receive epoetin beta at a starting dose of 2000 IU SC once weekly to reach and maintain a target Hb level of 10.5 to 11.5 g/dL. Standard treatment was as per investigator discretion.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta) | Total
Number analyzed (Participants) | 88 | 82 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (13.82) | 55.6 (12.64) | 56.2 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 45 | 41 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricle Mass Index (LVMI) at Month 15
Description: LVMI (in g/m^2) = (0.8 [1.04 {(LVEDD + IVS + PWT)^3 - (LVEDD)^3}] + 0.6) divided by BSA. Here, LVEDD = left ventricular end diastolic diameter (in centimeters [cm]); PWT = left ventricular posterior wall thickness in diastole (in cm); IVS = interventricular septal wall thickness in diastole (in cm). Echocardiogram was performed at baseline and Month 15 to interpret LVMI which was expressed in grams per meter square (g/m^2).
Time Frame: Baseline, Month 15
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Number analyzed (Participants) | 84 | 79
g/m^2 | 0.69 (26.34) | 0.10 (24.25)
Statistical Analysis 1: Comparison: Group 1 (Early Epoetin Beta) vs Group 2 (No/Late Epoetin Beta); Test type: Superiority or Other; p = 0.8811, ANCOVA with LOCF — P-value was calculated by ANCOVA with last observation carry forward (LOCF) method

2. Secondary Outcome: Left Ventricular End Systolic Volume Index (LVESVI)
Description: LVESVI was calculated by dividing left ventricular end systolic volume (LVESV) (in milliliters [mL]) with body surface area (BSA) (in meter square [m^2]). LVESVI is presented in milliliter per meter square (mL/m^2).
Time Frame: Baseline, Months 6 and 15
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome measure. Here "n"= participants who were evaluable for each category, for respective arm groups.
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Number analyzed (Participants) | 57 | 56
mL/m^2
  Baseline (n=57, 56) | 22.40 (6.36) | 21.04 (5.42)
  Month 6 (n=47, 53) | 26.86 (8.21) | 24.54 (8.06)
  Month 15 (n=54, 55) | 25.99 (9.31) | 25.03 (6.88)
Statistical Analysis 1: Comparison: Group 1 (Early Epoetin Beta) vs Group 2 (No/Late Epoetin Beta); Test type: Superiority or Other; p = 0.8864, ANCOVA with LOCF

3. Secondary Outcome: Left Ventricular End Diastolic Volume Index (LVEDVI)
Description: LVEDVI was calculated by dividing left ventricular end diastolic volume (LVEDV) (in mL) BSA (in m^2). LVEDVI was presented in mL/m^2.
Time Frame: Baseline, Months 6 and 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Number analyzed (Participants) | 57 | 56
mL/m^2
  Baseline (n=57, 56) | 61.08 (12.69) | 58.13 (10.83)
  Month 6 (n=47, 53) | 62.74 (15.41) | 60.40 (12.25)
  Month 15 (n=54, 55) | 62.26 (16.27) | 62.07 (11.36)
Statistical Analysis 1: Comparison: Group 1 (Early Epoetin Beta) vs Group 2 (No/Late Epoetin Beta); Test type: Superiority or Other; p = 0.5681, ANCOVA with LOCF

4. Secondary Outcome: Fractional Myocardial Shortening (FS)
Description: FS was calculated as: ([LVEDD - LVESD] divided by LVEDV) multiplied by 100; where LVEDD = left ventricular end diastolic diameter (in centimeters [cm]), LVESD = left ventricular end systolic diameter (in cm), LVEDV = left ventricular end diastolic volume (in mL). FS is expressed in percentage of LVEDV.
Time Frame: Baseline, Months 6 and 15
Population: ITT population. Here "n"= participants who were evaluable for each category, for respective arm groups.
Measure: Mean (Standard Deviation); unit: percentage of LVEDV
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Number analyzed (Participants) | 88 | 82
percentage of LVEDV
  Baseline (n=88, 82) | 36.45 (7.80) | 36.58 (8.97)
  Month 6 (n=84, 76) | 37.80 (7.40) | 38.49 (7.03)
  Month 15 (n=85, 79) | 37.58 (7.01) | 38.86 (7.52)
Statistical Analysis 1: Comparison: Group 1 (Early Epoetin Beta) vs Group 2 (No/Late Epoetin Beta); Test type: Superiority or Other; p = 0.1578, ANCOVA with LOCF

5. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF was calculated as ([LVEDV - LVESV], divided by LVEDV) multiplied by 100; where LVEDV = left ventricular end diastolic volume (in mL), LVESV = left ventricular end systolic volume (in mL). LVEF is expressed in percentage of LVEDV.
Time Frame: Baseline, Months 6 and 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of LVEDV
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Number analyzed (Participants) | 57 | 56
percentage of LVEDV
  Baseline (n=57, 56) | 63.44 (5.73) | 63.84 (5.44)
  Month 6 (n=47, 53) | 57.22 (6.87) | 59.92 (7.71)
  Month 15 (n=54, 55) | 58.63 (6.47) | 59.97 (6.46)
Statistical Analysis 1: Comparison: Group 1 (Early Epoetin Beta) vs Group 2 (No/Late Epoetin Beta); Test type: Superiority or Other; p = 0.2913, ANCOVA with LOCF

6. Secondary Outcome: Percentage of Participants With Stable Hb Levels Between 13 to 15 g/dL
Time Frame: Week 26 up to Week 64
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Number analyzed (Participants) | 86 | 81
percentage of participants | 75.6 [65.1 to 84.2] | 9.9 [4.4 to 18.5]
Statistical Analysis 1: Comparison: Group 1 (Early Epoetin Beta) vs Group 2 (No/Late Epoetin Beta); Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: up to 30 days after last study drug administration (35 months)
Arm/Group | Group 1 (Early Epoetin Beta) | Group 2 (No/Late Epoetin Beta)
Serious Adverse Events (participants affected / at risk) | 21/88 | 20/82
Other Adverse Events (participants affected / at risk) | 21/88 | 17/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Early Epoetin Beta) (N=88) | Group 2 (No/Late Epoetin Beta) (N=82)
Renal Impairment (Renal and urinary disorders) | 1 | 3
Renal failure chronic (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Perianal abscess (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Atherosclerosis (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Eye hemorrhage (Eye disorders) | 1 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 1
Generalized edema (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Early Epoetin Beta) (N=88) | Group 2 (No/Late Epoetin Beta) (N=82)
Hypertension (Vascular disorders) | 14 | 8
Edema peripheral (General disorders) | 8 | 9
Renal impairment (Renal and urinary disorders) | 5 | 4
Nasopharyngitis (Infections and infestations) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.